CLINICAL TRIAL: NCT01285713
Title: Effects of Glucose Containing Fluid in the Treatment of Acute Dehydration
Brief Title: IV Glucose for Dehydration Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: American Academy of Pediatrics (Other); Academic Pediatric Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-007632
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Results first posted 2013-01-23 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Dehydration
Keywords: Dehydration; Gastroenteritis; Dehydration in Gastroenteritis
MeSH Terms: conditions — Dehydration; Gastroenteritis | interventions — Glucose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5% Dextrose (D5) in Normal Saline (NS) (Experimental): 10cc/kg D5NS, followed by 30cc/kg NS
  Interventions: Drug: 5% Dextrose (D5) in Normal Saline (NS)
- Normal Saline (NS) (Active Comparator): 10cc/kg NS, followed by 30cc/kg NS
  Interventions: Drug: Normal Saline (NS)

INTERVENTIONS:
Drug: 5% Dextrose (D5) in Normal Saline (NS) — D5NS 10 cubic centimeter (cc)/kilogram (kg) to be followed by 30cc/kg of NS
  Other Names: D5NS
  Arms: 5% Dextrose (D5) in Normal Saline (NS)
Drug: Normal Saline (NS) — NS 10 cubic centimeter (cc)/kilogram (kg) to be followed by 30cc/kg NS
  Other Names: NS
  Arms: Normal Saline (NS)

SUMMARY:
To determine whether the addition of dextrose to IV fluids in the treatment of gastroenteritis leads to a decrease in serum ketones. Secondarily, the clinical benefits of dextrose containing fluids in the treatment of gastroenteritis will be assessed.

DETAILED DESCRIPTION:
Background: Evaluation and treatment of dehydration in gastroenteritis is a cornerstone of pediatric emergency medicine, however there are no standard regimens or guidelines for the amount or type of fluids administered when a child requires intravenous hydration. Reduced carbohydrate intake in gastroenteritis leads to free fatty acid breakdown, excess ketones, and an increased likelihood for continued nausea and vomiting. Glucose therapy can treat this catabolic metabolism, improving the ability to overcome dehydration and starvation, and facilitate a child's return to baseline. There has been no previous randomized controlled study examining the utility of early intravenous dextrose in the treatment of gastroenteritis.

Objectives: To determine whether the addition of dextrose to IV fluids in the treatment of gastroenteritis leads to a decrease in serum ketones. Secondarily, the clinical benefits of dextrose containing fluids in the treatment of gastroenteritis will be assessed.

Methods: This is a double blinded randomized controlled trial of children between the ages of 2 months and 12 years presenting to the Children's Hospital of Philadelphia (CHOP) Emergency Department (ED) who have gastroenteritis diagnosed by the ED attending or fellow and require intravenous hydration. Subjects will be randomized to either receive intravenous fluids containing dextrose or intravenous fluids without dextrose. The primary outcome measure is change in serum ketones during the intervention. Secondary outcomes are assessment of the clinical benefits of dextrose containing fluids in terms of persistence of emesis, satisfaction after treatment (physician and parental survey), admission rates, revisits within 1 week to the emergency department or to primary care physician, length of illness and parental assessment of time to return to baseline.

Implications: Despite our current standard of using normal saline for intravenous rehydration, there is a high admission rate with lengthy stays in the emergency department for children with gastroenteritis. There is room for improvement in the treatment of a very common emergency department entity. It is hypothesized that glucose load and subsequent increased endogenous insulin production will reduce free fatty acid breakdown and facilitate faster resolution of ketosis, and thus quicker return to baseline. By measuring serum ketones before and after intravenous fluid administration with either glucose or standard normal saline, we can directly measure these effects.

Inclusion Criteria

1. Males or females age 2 months to 12th birth date
2. Gastroenteritis (as diagnosed by ED attending or fellow physician)
3. Need for IV fluids
4. Dextrose stick of greater than 60 and less than 170
5. Parental/guardian English speaking and granting informed consent

Exclusion Criteria

1. Underlying chronic disease affecting glucose metabolism or reason/persistence of symptoms: Renal failure, Diabetes Mellitus, Diabetes Insipidus, Metabolic Disorder, ventriculoperitoneal (VP) shunt, Migraine Headaches
2. Shock
3. Vomiting greater than 72 hours since onset of illness
4. Patients that have received IV fluids at an outside institution within 12 hours

Investigational Plan: All enrolled subjects will have 1.5 microliters of blood collected onto a test strip during the IV placement performed for clinical care, and serum ketones will be measured using a bedside ketone meter. The ketone meter has been validated with comparison to standard laboratory beta-hydroxybutyrate levels (r=.92, p<0.0001). All patients will have a dehydration score recorded (Table 1). Subjects will be randomized to either the glucose containing IVF group or the non-glucose containing IVF group. All fluids will be prepared by a pharmacy and will be blinded to the treating team and patient. Those in the glucose containing IVF group will receive 10 cubic centimeter (cc) per kilogram (kg) (cc/kg) of 5%Dextrose (D5) in normal saline (NS)(D5NS) and then an 30 cc/kg bolus of normal saline. Those randomized to the non-glucose containing IVF group will receive 10 cc/kg of normal saline and then the rest of the normal saline bolus (30cc/kg). Both study arms will have the fluid intervention they initially received repeated once with the goal of a total of 40cc/kg to be completed within 60 minutes. D5NS was chosen to decrease the exposure to free water while suppressing lipolysis. After the intervention is complete, serum ketones will again be measured by bedside meter and recorded for all subjects. The treating team is blinded to the ketone measurements. A dextrose stick will be obtained with the final ketone measurement, and if the value is >200, the treating team will be notified to ensure proper safety. Subjects will not be allowed to have oral intake during this 60 minute study period in order to allow for determination of effect of intervention. A repeat dehydration score is obtained at time of disposition.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 2 months to 12th birth date
2. Gastroenteritis (as diagnosed by ED attending or fellow physician)
3. Need for IV fluids
4. Dextrose stick of greater than 60 and less than 170
5. Parental/guardian English speaking and granting informed consent

Exclusion Criteria:

1. Underlying chronic disease affecting glucose metabolism or reason/persistence of symptoms: Renal failure, Diabetes Mellitus, Diabetes Insipidus, Metabolic Disorder, VP shunt, Migraine Headaches
2. Shock
3. Vomiting greater than 72 hours since onset of illness
4. Patients that have received IV fluids at an outside institution within 12 hours

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Alpern, MD, Principal Investigator — Children's Hospital of Philadelphia; Kari Posner, MD, Principal Investigator — NYU Langone Health
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 5% Dextrose (D5) in Normal Saline (NS): 10cc/kg 5% Dextrose (D5) in Normal Saline (NS) (D5NS), followed by 30cc/kg Normal Saline (NS)
Period: Overall Study
Arm/Group | 5% Dextrose (D5) in Normal Saline (NS) | Normal Saline (NS)
Started | 42 | 41
Completed | 42 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- D5Normal Saline: 10cc/kg D5NS, followed by 30cc/kg NS
- Normal Saline: 10cc/kg NS, followed by 30cc/kg NS
- Total: Total of all reporting groups
Arm/Group | D5Normal Saline | Normal Saline | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 41 | 83
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.6 (3.3) | 3.4 (3.0) | 3.5 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 20 | 17 | 37
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 83

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Serum Ketones Before and After Administration of Intravenous Fluids for Acute Gastroenteritis
Description: Measurement of serum ketones by bedside ketone meter before and after administration of IVF for both groups to determine a change in serum ketones. The hypothesis is that dextrose containing IVF will lead to a decrease in serum ketones in children with acute gastroenteritis who require IV rehydration.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | D5Normal Saline | Normal Saline
Number analyzed (Participants) | 33 | 36
mmol/L | 1.10 (1.20) | 2.39 (1.62)
Statistical Analysis 1: Comparison: D5Normal Saline vs Normal Saline; Test type: Superiority or Other; p = 0.0003, Paired t-test

ADVERSE EVENTS:
Arm/Group | D5Normal Saline | Normal Saline
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 0/41 | 0/42

LIMITATIONS AND CAVEATS:
Single center study Small sample size Enrollment available 16 hours/day Evaluated one dextrose load of 500mg/kg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No